CLINICAL TRIAL: NCT02884765
Title: International, Multicenter, Prospective Registry to Collect Data of Treatment Patterns in Patients With Bilateral Condylar Fracture (BCFx) of the Mandible
Brief Title: Bilateral Condylar Fractures Registry
Acronym: BCFx
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AOCMF (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: RP_BCFx_1.0
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Bilateral Condylar Fracture of the Mandible
Keywords: mandibular condyle; subcondylar; mandible; fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bicondylar Fracture: Patients presenting a bilateral condylar fracture of the mandible with or without additional symphyseal fracture. Bilateral condylar fractures will be treated non-surgical, surgical or combining both.
  Interventions: Procedure: Non-surgical; Procedure: Non-surgical / Surgical; Procedure: Surgical

INTERVENTIONS:
Procedure: Non-surgical — Non-surgical treatment in both condylar fractures
Procedure: Non-surgical / Surgical — Non-surgical treatment in one condylar fracture and surgical treatment of the contralateral fracture
Procedure: Surgical — Surgical treatment in both condylar fractures

SUMMARY:
Prospective data will be collected in approximately 250 patients sustaining BCFx with or without any additional fracture(s) of the symphysis. Patients will be followed according to the standard (routine) at approximately 6 weeks and 3 months after the treatment. Data collection will include fracture details (i.e. classification, mechanism of injury), treatment details, functional and patient-reported outcomes, and anticipated or procedure-related adverse events (i.e. complications).

DETAILED DESCRIPTION:
Fractures of the condyles occur in around one third of patients sustaining a mandibular fracture. Bilateral fractures are reported in around one fifth to one third of all fractures of the mandibular condyles and are often combined with other fractures of the mandible or facial skeleton.

The treatment of condylar fractures, and in particular of bilateral condylar fractures (BCFx), is complex due to many different fracture patterns, surgeon's preferences, local constraints of the health care system and patient characteristics. Briefly, BCFx can be treated using either closed treatment (CTx) (e.g. intermaxillary fixation [IMF] and/or functional therapy) or surgical treatment (i.e. open reduction and internal fixation [ORIF]) in both fractures, or a combination of closed treatment and ORIF. The relationship of these treatments with the final outcome remains elusive, since the available literature does not report specific data for patients sustaining BCFx and has ignored or inadequately reported patient-reported outcomes. Consequently there is a lack of clinical evidence to assist the decision-making process.

Therefore, the purpose of this registry is to collect data in a standardized manner regarding the treatment, the clinical and the patient-oriented outcomes, and the complications of BCFx.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years at the time of the fracture
* Diagnosis of bilateral condylar fracture of the mandible with or without a concomitant fracture of the symphysis
* Dentition: Patients must have enough maxillary and mandibular teeth present to identify proper occlusion

Exclusion Criteria:

* Unilateral condylar fracture
* Additional maxillary fracture(s)
* Polytrauma (i.e. life threatening condition)
* Patients being treated with antiresorptive drugs at the time of inclusion or during their participation in the registry
* Pregnancy
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present registry

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients sustaining a bilateral condylar fracture of the mandible.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Mandibular movements (mobility index) | 3 months
  * Interincisal opening/maximal opening is defined as distance in millimeters between the edges of the incisors of the mandibular and the maxillary bone.
  * Lateral movements: With the mandible slightly open, it is defined as the distance in millimeters from the labioincisal embrasure between the central incisors to the labioincisal embrasure of the mandibular incisors
  * Protrusive movement: With the mandible slightly open, it is defined as the distance in millimeters between the incisal edges of the maxillary central incisor to the mandibular central incisor.
  Depending on the score, the mobility index will be calculated as follow:
  * 0 points: normal mandibular mobility
  * 1 - 4 points: slightly impaired mobility
  * 5 - 20 points: severely impaired mobility

OTHER OUTCOMES:
Mandible dysfunction (Helkimo Index) | 6 weeks / 3 months
Clinical evaluation of the occlusion status | 6 weeks / 3 months
  * Normal for the patient
  * Abnormal for the patient (anterior open bite / crossbite / lateral open bite in the premolar area / lateral open bite in the mola area)
Pain (numeric rating scale) | 6 weeks / 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ellis 3rd, DDS MS, Principal Investigator — University of Texas
Locations (21):
- United States (3):
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Helsinki University Hospital, Helsinki, Finland
- Germany (2):
  - Universitaetsklinikum Eppendorf, Hamburg
  - LMU - Klinikum der Universität München, Munich
- Hospital Sungai Buloh, Sungai Buloh, Malaysia
- Mexico (2):
  - Hospital General de Especialidades, Campeche
  - Hospital Trauma y Ortopedia Lomas Verdes, Mexico City
- Eramus MC, Rotterdam, Netherlands
- Mayo Hospital Lahore, Lahore, Pakistan
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- King Edward VIII Hospital, Durban, South Africa
- Spain (3):
  - Hospital Vall d' Hebron, Barcelona, Catalonia
  - 12 de Octubre University Hospital, Madrid
  - University Hospital La Paz de Madrid, Madrid
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Universitätsspital Zürich, Zurich
- National Cheng Kung University Hospital, Tainan, Taiwan
- Lviv Regional Clinical Hospital, Lviv, Ukraine
- Hospital Maciel de Montevideo, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No